CLINICAL TRIAL: NCT07400679
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, PARALLEL GROUP STUDY TO ASSESS RELATIVE BIOAVAILABILITY OF PF-08653944 WHEN ADMINISTERED ACROSS DIFFERENT INJECTION SITES IN ADULTS WITH OVERWEIGHT OR OBESITY
Brief Title: A Study to Learn How the Study Medicine Called PF-08653944 is Taken up Into the Blood in Adults With Overweight or Obesity.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C6491016
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Overweight; Obesity; Healthy
Keywords: Obesity; Overweight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment 1 (Experimental): Participants will receive a single subcutaneous (SC) dose of PF-08653944 on Day 1 administered to the abdomen.
  Interventions: Drug: PF-08653944
- Treatment 2 (Experimental): Participants will receive a single SC dose of PF-08653944 on Day 1 administered to the thigh.
  Interventions: Drug: PF-08653944
- Treatment 3 (Experimental): Participants will receive a single SC dose of PF-08653944 on Day 1 administered to the upper arm.
  Interventions: Drug: PF-08653944
- Treatment 4 (Optional) (Experimental): Japanese participants will receive a single SC dose of PF-08653944 on Day 1 administered to the abdomen.
  Interventions: Drug: PF-08653944

INTERVENTIONS:
Drug: PF-08653944 — Solution for injection
  Other Names: MET097

SUMMARY:
This study is being done to learn how the study medicine affects the body and how safe it is for people who take it. The researchers will look at a number of health tests, including blood tests such as calcitonin, amylase, and lipase, because similar medicines have sometimes caused changes in these tests.

This study is seeking participants who are:

* Adults who are obese or overweight with weight-related health conditions, and
* meet health and other checks assessed by the study doctor.

The study team will give a single dose of the study treatment at the clinic to the participants. At each study visit, blood samples will be collected, vital signs will be checked, and the study team will ask about any reactions or health changes. Vital signs are basic measurements that show how well the body is working. They help the study team quickly understand a participant's overall health. These usually include body temperature, heart rate, breathing rate, and blood pressure.

The study involves multiple clinic visits at a study site over the length of the study. The information collected will help researchers understand how the study medicine works and whether it is safe.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants 18 years of age or older at Screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECGs.
* BMI of 27-45 kg/m2 ; and a total body weight >50 kg (110 lb).
* For Japanese participants only: BMI of 20-45 kg/m2 and a total body weight >50 kg (110 lb) and must have 4 biological Japanese grandparents who were born in Japan.

Key Exclusion Criteria:

* Pregnant or breastfeeding women, or those planning pregnancy during the study.
* Clinically significant medical conditions including hematologic, renal, endocrine, pulmonary, gastrointestinal (including pancreatitis, gallbladder disease, clinically relevant gastric emptying disorders), cardiovascular, hepatic, psychiatric, neurologic, or severe allergic diseases.
* Personal or first-degree family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2), or suspected MTC.
* Active or recent suicidal ideation in the past year, suicidal behavior within the past 5 years, or any psychiatric condition that increases risk in the investigator's judgment.
* Clinically significant gastric emptying abnormality or chronically taking drugs that directly affect GI motility.
* Acute gastrointestinal symptoms at screening or Day -1.
* Known hypersensitivity to PF-08653944, GLP-1 receptor agonists, or any excipients.
* Prior participation in any study involving PF-08653944 (formerly MET097) with at least one dose received.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of PF-08653944 | Up to 85 days
  To assess the relative bioavailability of SC to the thigh or upper arm compared to the abdomen
PK: Maximum Observed Concentration (Cmax) of PF-08653944 | Up to 85 days
  To assess the relative bioavailability of SC to the thigh or upper arm compared to the abdomen

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 85 Days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.